CLINICAL TRIAL: NCT07273721
Title: Efficacy and Safety of BT200 (Rondoraptivon Pegol) in Patients With Type 2B Von Willebrand Disease
Brief Title: Efficacy and Safety of BT200 (Rondaptivon Pegol) in Patients With Type 2B Von Willebrand Disease
Acronym: BT200-VWD2B
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Schoergenhofer, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT200-VWD2B Version 1.1; 2024-518294-34-01 (EU CTIS Number)
Record Dates: First submitted 2025-09-29; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Von Willebrand Disease (VWD), Type 2
Keywords: von Willebrand's disease; thrombocytopenia; bleeding; placebo
MeSH Terms: conditions — von Willebrand Diseases; Thrombocytopenia; Hemorrhage

STUDY DESIGN:
Intervention Model Description: randomized, controlled, double blind, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo is non-distinguishable from verum based on physicochemical properties (colourless fluid)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients randomized to receive placebo first. They will receive the verum BT200 after an adequate washout period
  Interventions: Drug: Placebo
- BT200 (Experimental): Patients randomized to receive BT200 (verum) first and placebo in the second phase after an adequate washout period.
  Interventions: Drug: BT200

INTERVENTIONS:
Drug: BT200 — Aptamer directed against the A1 domain of von Willebrand factor
  Arms: BT200
Drug: Placebo — Placebo for BT200
  Arms: Placebo

SUMMARY:
This randomized clinical trial with a cross-over design is being conducted at the Department of Clinical Pharmacology at the Medical University of Vienna, and a total of 4-6 patients with type 2B von Willebrand disease (VWD) will participate.

The main purpose of this clinical trial is to investigate the efficacy and safety of BT200, a new drug for thrombocytopenic patients with type 2B von Willebrand disease (VWD). Based on previous studies, we expect that this drug will inhibit the breakdown of von Willebrand factor (VWF) in small doses, leading to an increase in von Willebrand factor (VWF), platelet count, and factor VIII. This should also lead to a reduced tendency to bleed.

This study will begin with an observation phase and will then proceed in two periods of approximately 64 days each:

Placebo or BT200 will be administered subcutaneously at a dose of 12 mg on the first day of the study. After that, patients will self-administer the drug at a dose of 6 mg (0.4 mL) or placebo once a week for another 4 weeks starting the following week (a total of 4 times over a period of 4 weeks). During this time, they will be asked to come to our clinic for a follow-up visit.

After a "washout phase" lasting several weeks, during which patients do not receive the study drug/placebo but are asked to record any bleeding events, the second period begins on day 64:

BT200 or placebo is administered again, depending on what the patients received in the first period. Patients therefore receive the study drug for 4 weeks and placebo for 4 weeks; which is administered when is randomized; a follow-up examination also takes place during this period.

At the end of the second period, there is another "washout phase" lasting several weeks. On day 127, the final examination takes place at the clinic, after which patients have the opportunity to participate in an extension study (to be amended).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Type 2B VWD with thrombocytopenia and a recent bleeding history (e.g. recurrent haematomas)
3. Able to comprehend and to give informed consent
4. Able to cooperate with the Investigator, to comply with the requirements of the study, and to complete the full sequence of protocol-related procedures

Exclusion Criteria:

1. Clinically significant medical history or ongoing chronic illness that would jeopardise the safety of the patient or compromise the quality of the data derived from his/her participation in this study
2. History of significant drug allergy or anaphylactic reactions
3. Substance abuse, mental illness, or any reason that makes it unlikely in the judgment of the Investigator for the patient to be able to comply fully with study procedures
4. Use of medication during 2 weeks before the start of the study, which in the judgment of the Investigator may adversely affect the patient's welfare or the integrity of the study's results
5. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days or 5 elimination half-lives (whichever is longer) prior to treatment start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome measure Platelet Counts | During the five-week Treatment Phase compared with the five-week Control Phase
  Platelet Counts
Co-Primary Endpoint Clinically evident bleeding | During the five-week Treatment Phase compared with the five-week Control Phase
  number of clinically evident bleedings

SECONDARY OUTCOMES:
von Willebrand factor antigen | During the five-week Treatment Phase compared with the five-week Control Phase
  Concentration of von Willebrand factor antigen quantified by Enzyme-linked immunoassay
von Willebrand factor activity | During the five-week Treatment Phase compared with the five-week Control Phase
  von Willebrand factor activity quantified by Gp1bM assay
VWF activity collagen binding | During the five-week Treatment Phase compared with the five-week Control Phase
  Activity of VWF quantified with a collagen binding assay
VWF:ristocetin co-factor activity | During the five-week Treatment Phase compared with the five-week Control Phase
  Activity of VWF quantified with a ristocetin co-factor assay
Enzyme-linked immunosorbent assay (ELISA) for unbound VWF-A1 domain (REAADS® ) | During the five-week Treatment Phase compared with the five-week Control Phase
  Concentration of unbound VWF-A1 domain quantified by Enzyme-linked immunosorbent assay (ELISA) (REAADS® )
Platelet function under high shear rates | During the five-week Treatment Phase compared with the five-week Control Phase
  Platelet Function Analyzer
BT200 plasma concentrations | During the five-week Treatment Phase compared with the five-week Control Phase
  plasma concentrations of BT200
Serious, drug-related AEs | During the five-week Treatment Phase compared with the five-week Control Phase
  Serious, drug-related AEs
Premature terminations due to drug-related AEs | During the five-week Treatment Phase compared with the five-week Control Phase
  Number of participants who premature terminate treatment due to drug-related AEs
Adverse events indicative of BT200 toxicity | During the five-week Treatment Phase compared with the five-week Control Phase
  Patterns of serious or non-serious, drug-related AEs, and/or clinically relevant laboratory abnormalities, vital signs, or physical findings suggestive of one or more specific target organs for toxicity of BT200

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request to the PI.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Publication of the trial results, within 3 months of reasonable request to the PI
Access Criteria: Fellow Researchers with a reasonable proposal for planned analyses may contact the PI. Anonymized individual data may be shared.